CLINICAL TRIAL: NCT06214143
Title: A Single-arm, Multi-center Phase Ib/IIa Clinical Study to Evaluate the Tolerability, Safety, and Initial Efficacy of T3011 Herpesvirus Injection Combined With PD-1/PD-L1 Inhibitors in Patients With Advanced Solid Tumors
Brief Title: A Clinical Study of T3011 in Combination With PD-1/PD-L1 Inhibitors in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH-T3011-201
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T3011 (Experimental)
  Interventions: Biological: T3011 high dose; Biological: T3011 middle dose; Biological: T3011 low dose

INTERVENTIONS:
Biological: T3011 high dose — T3011 high dose： T3011 will be given intratumorally，Q2W； PD-1/PD-L1 inhibitor：Administered by intravenous infusion，3 mg/kg，Q2W
Biological: T3011 middle dose — T3011 middle dose： T3011 will be given intratumorally，Q2W； PD-1/PD-L1 inhibitor：Administered by intravenous infusion，3 mg/kg，Q2W
Biological: T3011 low dose — T3011 low dose： T3011 will be given intratumorally，Q2W； PD-1/PD-L1 inhibitor：Administered by intravenous infusion，3 mg/kg，Q2W

SUMMARY:
This clinical study evaluated the efficacy and safety of T3011 in combination with PD-1/PD-L1 inhibitors in subjects with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with advanced solid tumors;
2. At least one measurable lesion;
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
4. Expected survival > 12 weeks;
5. Laboratory inspection meets the requirements;
6. For women of childbearing potential, the serum pregnancy test results must be negative prior to the first dose，and effective contraceptive measures must be taken from signing the informed consent form (ICF) until at least 6 months after the last dose;
7. Male subjects of childbearing potential agree to use effective contraception from signing the ICF until at least 6 months after the last dose; In addition, male subjects must agree not to donate sperm during this period;
8. Understand and voluntarily sign the ICF，willing and able to comply with all experimental requirements.

Exclusion Criteria:

1. Subjects who have received other antitumor therapy within the prescribed time prior to the first dose;
2. Subjects with a history of other malignancies within the prescribed time prior to the start of study treatment.
3. At screening, subjects with a history or evidence of high risk cardiovascular disease;
4. Subjects with persistent or active infection requiring intravenous anti-infective therapy;
5. Subjects with autoimmune diseases or a history of autoimmune diseases;
6. Subjects with known psychiatric disorders that may affect trial compliance;
7. Subjects who have pleural effusion, pericardial effusion, or ascites before starting treatment and require puncture drainage, or who had received puncture drainage within the specified time before starting the study treatment;
8. Subjects requiring systemic treatment with anti-HSV drugs during the study period;
9. Subjects who have received live or attenuated vaccines within the prescribed time prior to the first dose, or who plan to receive such vaccines during the study period; Subjects who have received any tumor vaccine in the past;
10. Subjects who had undergone major surgery within the prescribed time before the first dose，and had not recovered from surgery-related adverse reactions or were still in the postoperative recovery period，or who plan to undergo major surgery during the study period;
11. Subjects with a history of drug use，drug abuse or alcohol abuse within the year prior to signing the ICF;
12. Female subjects who are pregnant or breastfeeding, or planning to conceive or have children during the study period;
13. The investigator considers it inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Approximately 2years
  Adverse event type, incidence, duration
Objective response rate(ORR) | Approximately 2years
  Tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | Approximately 2years
  DCR was defined as the percentage of patients who have achieved complete response, partial response and stable disease
Duration of remission (DOR) | Approximately 2years
  DOR was defined for participants who had an objective response as the time from the first occurrence of a documented unconfirmed response to the date of disease progression per RECIST v1.1 or death from any cause.
Progression-free survival (PFS) | Approximately 2years
  From the start date of study treatment to the date of progression disease or death , whichever occurred first.
Overall Survival (OS) | Approximately 2years
  Determination of the overall survival time of all patients

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Anyang Cancer Hospital, Anyang
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - Hunan cancer hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - Dongguan People's Hospital, Dongwan
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Harbin Medical University Cancer Hospital, Ha’erbin
  - Shandong cancer hospital, Jinan
  - Jiangxi cancer hospital, Nanchang
  - Guangxi Medical University Affiliated Cancer Hospital, Nanning
  - Shanghai East Hospital, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai
  - Liaoning Cancer Hospital, Shenyang
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen
  - Shanxi Cancer Hospital, Taiyuan
  - Tianjin cancer hospital, Tianjin
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Henan cancer hospital, Zhengzhou